CLINICAL TRIAL: NCT05259215
Title: Predicting Independent Walking Ability Using the Simplified Stroke Rehabilitation Assessment of Movement, Berg Balance Scale, Barthel Index for Activities of Daily Living in Individuals Post Stroke: an Observational Pilot Study
Brief Title: Predicting Independent Walking Ability Using the Simplified Stroke Rehabilitation Assessment of Movement, Berg Balance Scale, Barthel Index for Activities of Daily Living in Individuals Post Stroke
Status: Completed | Type: Observational
Sponsor: Ukrainian Association of Physical Therapy (Other)
Responsible Party: Principal Investigator, Mykola Romanyshyn, Senior physiotherapist, Ukrainian Association of Physical Therapy
Other Study IDs: UAPT 0001
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-walking group
  Interventions: Other: physiotherapy
- independently walking group
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — Standard usual care physiotherapy after stroke

SUMMARY:
Cohort observational retrospective pilot study by design. The purpose of this study was to determine a cut scores to predict independent ambulation for the Simplified Stroke Rehabilitation Assessment of Movement, Berg Balance Scale, Barthel Index for Activities of Daily Living.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with stroke after the age of 17 confirmed stroke by neuroimaging, understanding instructions, time after stroke up to 1 year.

Exclusion Criteria:

* Subjects were excluded if they have: the presence of aphasia that would have interfered with the participant's ability to understand and comply with study procedures or complete stroke assessments, dementia, ataxia, localization of stroke in the cerebellum or vertebrobasilar insufficiency, orthopedic problems that affected the ability to walk before the stroke and time after stroke more than 1 year.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with stroke
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Category | 1-5 minutes
  The Functional Ambulation Categories (FAC) is a 6-point functional walking test that evaluates ambulation ability, determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.

SECONDARY OUTCOMES:
Simplified Stroke Rehabilitation Assessment of Movement (S-STREAM) | 15-20 minutes
  The Stroke Rehabilitation Assessment of Movement (STREAM) instrument was designed to provide a comprehensive and quantitative evaluation of voluntary movements (ie, an impairment measurement) and basic mobility (ie, a disability measurement) in patients with stroke.
Berg Balance Scale (BBS) | 15-20 minutes
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Barthel Index for Activities of Daily Living (BI) | 15-20 minutes
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.

CONTACTS AND LOCATIONS:
Locations (1):
- communal non-commercial enterprise "Kyiv Regional Clinical Hospital", Department of Rehabilitation of Patients with Consequences of Diseases and Injuries of the Nervous System, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No